CLINICAL TRIAL: NCT00205985
Title: Comparison of Time to Return to Previous Activity Between Operative Treatment and Cast Immobilization of Complete Fracture of the Middle Part of the Scaphoid Without Dislocation
Brief Title: Operative Versus Conservative Treatment of Scaphoid Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Organization: AO Innovation Translation Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-scaph-04
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Scaphoid Fracture
Keywords: Return to work; Scaphoid fracture; Operative treatment; Activity level

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Scaphoid screw — Conservative treatment versus application of scaphoid screw

SUMMARY:
The aim of this study is to compare the time to return to previous activity

level between operative treatment and non-operative cast immobilization of

patients with an acute complete fracture of the middle part of the scaphoid,

without any dislocation or comminution visible CT-scan.

ELIGIBILITY:
Inclusion Criteria:

* Mature skeleton
* Isolated, acute complete fracture of the mid third of the scaphoid

Exclusion Criteria:

* acute fractures of both hands
* one hand missing
* other injuries than scaphoid fractures
* rheumatoid, osteoarthritis or polyarthritis
* previous soft tissue injuries of the hand
* drug or alcohol abuse
* participant in trial during the previous month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-12; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Time to return to previous activity level
Time to return to full work and household duties

SECONDARY OUTCOMES:
DASH
SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schaedel-Hoepfner, Prof. MD, Principal Investigator — Klinikum der Universitaet Marburg
Locations (1):
- Klinikum der Philipps Universitaet Marburg, Marburg, Germany

REFERENCES:
- [Result] Pfeiffer BM, Nubling M, Siebert HR, Schadel-Hopfner M. A prospective multi-center cohort study of acute non-displaced fractures of the scaphoid: operative versus non-operative treatment [NCT00205985]. BMC Musculoskelet Disord. 2006 May 11;7:41. doi: 10.1186/1471-2474-7-41. PMID 16689987